CLINICAL TRIAL: NCT06849908
Title: A Multi-center, Prospective, Open-label, Randomized Study to Explore Efficacy and Safety of Baricitinib in Refractory Intestinal Behçet's Syndrome Patients
Brief Title: Baricitinib in the Treatment of Intestinal Behçet's Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Baricitinib-IBS-PUMCH
Record Dates: First submitted 2024-07-31; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Behcet Syndrome, Intestinal Type
Keywords: Baricitinib; Adalimumab; Intestinal Behçet's Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — baricitinib; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baricitinib for IBS (Experimental)
  Interventions: Drug: Baricitinib
- Adalimumab for IBS (Experimental)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Baricitinib — Participants randomized to this arm will maintain their original steroids and/or immunomodulators, combined with Baricitinib 4 mg/day for 6 months.
  Other Names: Olumiant®
  Arms: Baricitinib for IBS
Drug: Adalimumab — Participants randomized to this arm will maintain their original steroids and/or immunomodulators, combined with ADA (initially ADA 160 mg subcutaneous injection, followed by 80 mg ADA after 2 weeks, then 40 mg ADA every 2 weeks thereafter) for 6 months.
  Other Names: Humira®
  Arms: Adalimumab for IBS

SUMMARY:
This study aims to conduct a randomized controlled trial to compare the efficacy and safety of Baricitinib and Adalimumab (ADA) in the treatment of refractory intestinal Behçet's Syndrome (BS). The objective is to demonstrate if Baricitinib is non-inferior to ADA in controlling BS inflammation, reducing BS recurrence， alleviating gastrointestinal symptoms and promoting intestinal mucosal healing.

DETAILED DESCRIPTION:
The non-inferiority will be established by comparing the lower bound of the two-sided 95% confidence interval with the non-inferiority margin. If the lower bound was larger than the margin, Baricitinib would be regarded as non-inferiror to ADA. Superority will be further assessed in case that the non-inferiority is established. Both ITT and PP analysis will be conducted for the primary outcome given the non-inferiority design. Trial result will be primarily interpreted based on ITT analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Refer to the consensus on the diagnosis and treatment of intestinal Behçet's syndrome in China: Patients who meet the 2013 International Criteria for Behçet's Disease (ICBD) and have typical Behçet's syndrome-related intestinal ulcers confirmed by colonoscopy, or patients diagnosed according to the criteria for Behçet's syndrome established by the Korean Behçet's Disease Collaborative Group in 2009;
2. Patients have a DAIBD score ≥ 40 points or intestinal symptom score ≥ 3 points at baseline;
3. Endoscopic examination conducted within 60 days before inclusion suggests active intestinal ulcers;
4. Patients who have been treated with medium to high-dose steroids (prednisolone equivalent of 0.5-1 mg/kg/day) for more than 1 month continuously, or any immunomodulator/Immunosuppressants for more than 3 months regularly or biologics for more than 2 months, as judged by the doctor to be treatment failure or intolerance;
5. Currently steroid dose ≤ 30 mg prednisolone equivalent, stabilized for ≥ 2 weeks, and/or stabilized immunomodulator dose for ≥ 4 weeks;
6. Understanding the research process, voluntary participation, and signing of informed consent.

Exclusion Criteria:

1. Diagnosis of other diseases such as Crohn's disease, ulcerative colitis, lymphoma, etc.;
2. Other active organ damage related to BS requires intensified immunosuppressive therapy, including aneurysms, uveitis, and substantial involvement of the central nervous system; skin lesions and joint involvement can be included;
3. Severe organ dysfunction including ALT, AST, TBIL levels exceeding twice the upper limit of normal, creatinine levels exceeding 1.5 times the upper limit of normal, white blood cell count < 3×10^9/L, ANC < 2×10^9/L, hemoglobin < 80g/L, platelets < 100×10^9/L;
4. Active infections such as active tuberculosis, active hepatitis B or C, syphilis, chronic Epstein-Barr virus infection, HIV infection, sustained or severe bacterial or viral infections, and history of severe herpes zoster;
5. Patients with latent tuberculosis must undergo ≥3 weeks of prophylactic anti-tuberculosis treatment before inclusion;
6. Primary immunodeficiency disease;
7. History of cancer, or endoscopic intestinal histopathology indicating intraepithelial neoplasia or malignancy, or presence of other malignancies;
8. Patients who did not respond to infliximab treatment for primary refractory BS (patients with secondary failure, intolerance, or allergy to infliximab should be included);
9. Patients treated with biologics/small molecule targeting therapies within 5 half-lives (including use of tofacitinib within 10 days, etanercept within 4 weeks, infliximab within 8 weeks, golimumab, certolizumab, abatacept, and tocilizumab within 10 weeks, ustekinumab within 6 months);
10. Patients with prior use of baricitinib or ADA;
11. Complications of intestinal BS such as symptomatic stenosis, short bowel syndrome, intestinal fistula, or suspected intra-abdominal abscess; potential need for surgery or situations not conducive to DAIBD and efficacy assessment; any form of intestinal resection or other abdominal surgery within 6 months before baseline; presence of a functioning (i.e., patent) stoma or ostomy;
12. Patients requiring parenteral nutrition due to disease severity;
13. Pregnant, lactating, or planning pregnancy soon;
14. Patients unwilling or unable to comply with regular visits;
15. History of severe thrombotic events or chronic cardiovascular events.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with marked improvement (MI) at week 24 of follow-up | Baseline to week 24
  Based on the combined assessment of gastrointestinal symptoms and endoscopy scores[1], gastrointestinal symptom scoring is defined as follows: 0 points, asymptomatic; 1 point, does not affect daily life; 2 points, mildly affects daily life; 3 points, moderately affects daily life; 4 points, severely affects daily life. Endoscopy scoring is defined as follows: 0 points, mucosal healing; 1 point, maximum ulcer ≤ original 1/4; 2 points, maximum ulcer between original 1/4 and 1/2; 3 points, maximum ulcer ≥ original 1/2 or enlargement. Marked improvement is defined as gastrointestinal symptom and endoscopy scores both ≤ 1.
  [1]Sugimura, N. et al. Real-world efficacy of adalimumab and infliximab for refractory intestinal Behçet's disease. Dig. Liver Dis. 51, 967-971 (2019).

SECONDARY OUTCOMES:
Proportion of patients with CR (complete response) at week 24 of follow-up | Baseline to week 24
  CR is defined as both gastrointestinal symptoms and endoscopy scores being 0.
Proportion of patients with improvement of ≥1 point in gastrointestinal symptom scores compared to baseline at week 24 of follow-up | Baseline to week 24
Changes in C-reactive protein (CRP) compared to baseline | Baseline to week 24
  The hs-CRP is acute phase reactants that are indicative of the patient's disease activity.
Changes in erythrocyte sedimentation rate (ESR) compared to baseline | Baseline to week 24
  The ESR is acute phase reactants that are indicative of the patient's disease activity.
Changes in DAIBD scores compared to baseline | Baseline to week 24
  Disease Activity Index for Intestinal Behcet's Disease (DAIBD)；
Changes in BDCAF scores compared to baseline | Baseline to week 24
  Behçet's Disease Current Activity Index (BDCAF)；
Changes in SF-36 of life questionnaires compared to baseline | Baseline to week 24
  Short Form (36) Health Survey(SF-36);
Changes in IBDQ quality of life questionnaires compared to baseline | Baseline to week 24
  Inflammatory Bowel Disease Questionnaire (IBDQ)
Incidence of Treatment-Emergent Adverse Events | Baseline to week 24
  Record the types, frequency, and severity of adverse events, as well as the number of study participants who were drop out due to any adverse events. Adverse event: Any medical condition that affects the health of the participant during the study or worsens a preexisting medical condition, regardless of whether it is causally related to the study, is considered an adverse event.
  This can be symptoms, signs, or abnormal laboratory tests. Serious adverse event (SAE): Any significant medical event that causes death, is life-threatening, requires hospitalization, results in permanent or severe disability or loss of function, or the investigator deems it a significant medical event that may seriously harm the participant or require medical intervention to prevent the above outcomes.
  The causal relationship between the serious adverse event and the study is determined by the investigator's discussion.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No